CLINICAL TRIAL: NCT02861274
Title: ELectrophysiological Mechanisms Underlying the Inhibitory CArdiac Syncope: Therapeutic and Prognostic Implications The ELICA Study
Brief Title: Electrophysiological Mechanisms and Inhibitory Cardiac Syncope
Acronym: ELICA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Celestino Sardu, MD, MSc, PHD, University of Campania Luigi Vanvitelli
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 7.2016
Record Dates: First submitted 2016-08-01; First posted 2016-08-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Syncope Recurrent

ARMS (2):
- electrophysiological testing (Active Comparator): Patients will receive a pacemaker.
  Interventions: Device: pacemaker
- control group (No Intervention): These subjects will receive cardicor® (beta blockers).

INTERVENTIONS:
Device: pacemaker
  Arms: electrophysiological testing

SUMMARY:
OBJECTIVES: To evaluate syncope recurrence at follow up in patients with a positive cardio inhibitory response to the head up tilt testing (HUT) evaluation.

METHODS: 36 consecutive patients affected by cardio inhibitory syncope to HUT without asystolia (2A type) have been enrolled in this study. These patients have been studied by electrophysiological study (ES). After ES patients have been differently treated (interventional treatment group A, v/s drug therapy group), and followed up during 360 days, to evaluate syncope recurrences.

ELIGIBILITY:
Inclusion Criteria:

* age more than 18, normal heart function, more than 1 syncope event for year.

Exclusion Criteria:

* age inferior 18 years, history of myocardial infarction, heart failure, structural heart disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-01; Primary Completion 2015-01 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
syncope recurrence | 360 days

REFERENCES:
- [Derived] Sardu C, Marfella R, Testa G, Santamaria M, Sacra C, Ranauro A, Paolisso G, Rizzo MR, Barbieri M. ELectrophysiological mechanisms underlying the Inhibitory CArdiac syncope without asystolic significant pause: Therapeutic and prognostic implications. The ELICA randomized trial. Medicine (Baltimore). 2018 Aug;97(31):e11757. doi: 10.1097/MD.0000000000011757. PMID 30075596